CLINICAL TRIAL: NCT05182203
Title: Safety and Retention Rate of the JAK and TNF Inhibitors in Rheumatoid Arthritis: a Real-life Experience
Status: Completed | Type: Observational
Sponsor: Tuen Mun Hospital (Other Government)
Responsible Party: Principal Investigator, Chi Chiu Mok, Consultant, Tuen Mun Hospital
Other Study IDs: HKSRJAK study
Record Dates: First submitted 2021-12-18; First posted 2022-01-10 (Actual); Last update posted 2023-02-22 (Actual); Status verified 2023-02

CONDITIONS: Rheumatoid Arthritis; Drug Use
Keywords: rheumatoid arthitis; biological agents; targeted agents
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Biological Products

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- JAK inhibitors: RA patients treated with JAK inhibitors
  Interventions: Drug: biologic/targeted therapy
- TNF inhibitors: RA patients treated with TNF inhibitors
  Interventions: Drug: biologic/targeted therapy

INTERVENTIONS:
Drug: biologic/targeted therapy — TNF inhibitors or the JAK inhibitors

SUMMARY:
This study aims to extract data from the Hong Kong Biologics Registry for retention rate of the JAK inhibitors in rheumatoid arthritis and review other adverse events by looking at the medical record retrospectively. These real life data are important as they cannot be provided by randomized controlled trials which are limited by the duration of observation and fixed protocols in research settings. Moreover, data will represent our local experience of the JAK inhibitors in Chinese patients with RA. The retention rate and adverse effects of the JAK inhibitors are compared with conventional TNF inhibitors.

DETAILED DESCRIPTION:
This study aims to extract data from the Hong Kong Biologics Registry for retention rate of the JAK inhibitors in rheumatoid arthritis and review other adverse events by looking at the medical record retrospectively. Efficacy data and adverse events, in particular major adverse cardiovascular events (MACEs) and malignancy will be looked at and compared with the TNF inhibitors. Retention / withdrawal rates of the drugs will be studied by statistical analyses.

ELIGIBILITY:
Inclusion Criteria:

* All RA patients in our biologics registry treated with the JAK inhibitors (N=411)
* All RA patients in our biologics registry treated with the TNF inhibitors (N=1392)

Exclusion Criteria:

- RA patients in our biologics registry treated with other biologic/targeted DMARDs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Diagnosis of RA Ever received treatment with any biologic/targeted DMARDs data entered into our Biologics registry age >=18 years
Sampling Method: Non-Probability Sample
Enrollment: 1732 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2022-10-01 (Actual)

PRIMARY OUTCOMES:
Withdrawal rate due to major / serious adverse events | from start of biologic/targeted DMARD use to these event(s) up to 10 years
  adverse events eg. MACEs, malignancy, infections

SECONDARY OUTCOMES:
Withdrawal rate due to inefficacy | from start of biologic/targeted DMARD use to last clinic visit up to 10 years
  Efficacy of the agents in terms of retention rate

CONTACTS AND LOCATIONS:
Overall Officials: Chi Chiu Mok, MD, FRCP, Principal Investigator — Tuen Mun Hospital
Locations (1):
- Department of Medicine, Tuen Mun Hospital, Hong Kong, China

IPD SHARING:
Plan to Share IPD: No